CLINICAL TRIAL: NCT01071395
Title: Validation of Dyskinesia Rating Scales
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Principal Investigator, Christopher G. Goetz, MD, MD, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: Valid Dyskin Rating Scales
Record Dates: First submitted 2010-02-17; First posted 2010-02-19 (Estimated); Results first posted 2015-05-28 (Estimated); Last update posted 2022-12-29 (Actual); Status verified 2022-11

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Dyskinesia; Dyskinesia Rating Scales; Amantadine; Placebo
MeSH Terms: conditions — Parkinson Disease; Dyskinesias | interventions — Amantadine; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Amantadine (Experimental): Amantadine 100mg tab BID or TID for duration of study
  Interventions: Drug: Amantadine
- Placebo (Placebo Comparator): Placebo one tab BID or TID for duration of study
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Amantadine — Amantadine hydrochloride 300mg daily in three divided doses
  Other Names: Symmetrel
  Arms: Amantadine
Drug: Placebo — Sugar pill given 3 times daily
  Other Names: sugar pill
  Arms: Placebo

SUMMARY:
This study will evaluate the responsiveness of a variety of available dyskinesia rating scales to treatment with amantadine or placebo in Parkinson's disease patients with dyskinesia. The study will be a parallel, double-blind, randomized trial of 68 patients treated with amantadine or placebo for 8 weeks. Pre-treatment evaluations will be performed and compared to end of study evaluations on the best treatment dose (200 or 300 mg amantadine or matching placebo) daily. Safety evaluations will be conducted.

The responsiveness of the different scales will be evaluated statistically with a mixed model in which changes in the outcome measures over time will include a fixed effect of treatment group assignment. The model will additionally account for random effects of intercepts (the scale scores at baseline) that will include both random variation (person-specific) and specific variation associated with rate of change in outcome. The investigators may include adjustments for possible confounding covariates, including baseline demographics and center. The goal of the program is to provide researchers with the best scale(s) to distinguish dyskinesia change in Parkinson's disease (PD) associated with amantadine in comparison to placebo and to establish the magnitude of effect achievable with amantadine as a comparator "gold standard" that must be met or surpassed by future anti-dyskinetic agents. Additionally, with the use of paper and pencil questionnaires, the study will investigate the impact of patient optimism and patient and rater expectation of positive effects on the dyskinesia rating outcomes.

DETAILED DESCRIPTION:
Objective/Rationale:

Dyskinesias, or involuntary jerking movements, are troublesome problems for many Parkinson's disease patients. Chemical studies have led to the development of several new treatment strategies. However, because dyskinesias are cause various degrees of difficulty for patients and are often perceived by patients and caregivers differently than by doctors, the rating of dyskinesias remains a scientific challenge. This program will examine a wide gamut of available rating scales to determine which one(s) detect change during dyskinesia treatment. Establishing excellent measurement tools of dyskinesias will allow future treatments to be evaluated in a uniform and maximally effective manner.

Project Description:

An team of experts will test several dyskinesia scales in a group of Parkinson's disease patients with dyskinesia. Patients will be treated with either amantadine or placebo (an inactive product). The study will be "blinded" so that the raters and the patients do not know if a given patient is receiving amantadine or placebo. Amantadine is selected for this trial, because it is the only drug that has received the designation of Efficacious for dyskinesia by the Movement Disorder Society. This conclusion was based however, on small studies and no large clinical trial of this drug has been conducted in dyskinetic patients. The scales will assess dyskinesia before and after several weeks of treatment.

Relevance to Diagnosis/Treatment of Parkinson's Disease:

This study will establish a "gold standard" for rating dyskinesia in future trials of treatments in Parkinson's disease patients. It will allow physicians to know the level of change that occurs with a standard and available treatment (amantadine) and to compare that level with changes that occur with newer treatments. Patients will benefit from this new international standard, because they can compare the likelihood and magnitude of anticipated improvement from different dyskinesia treatments, whether medical or surgical.

Anticipated Outcome:

The anticipated outcomes of this study are:

* The impact of amantadine treatment on dyskinesia will be clearly defined.
* The effect that participation in a clinical program, even if no amantadine is given ("placebo improvements") will be delineated.
* A hierarchy of numerous scales will be determined based on their absolute and relative capability to detect change during treatment.
* The best scale(s) to evaluate dyskinesia in clinical practice and research efforts will be identified.

ELIGIBILITY:
Inclusion Criteria:

1. Parkinson's disease patient, defined by United Kingdom Brain Bank criteria
2. Current age between 30-90
3. Clinically pertinent dyskinesias defined by Clinical Gl;obal Impression-severity score (see attachment) > 3 (mild) established by clinician's total assessment of patient including objective observation during the screening process. *
4. Documentation of creatinine level at screening evaluation that is within the normal range for the local university laboratory.
5. Stable doses of all antiparkinsonian medications for at least 4 weeks
6. No treatment with amantadine for at least 3 months.
7. Presence of a caregiver willing to participate in the study
8. Subjects/caregivers must demonstrate the capacity to complete an accurate home diary based on training and evaluation during the screening period (see attached training rules).
9. Subjects must be able to provide written informed consent.
10. If the subject received amantadine in the past, the drug was stopped for reason other than adverse events.
11. In the opinion of the enrolling investigator, the subject will be able to maintain current dosing schedule of antiparkinsonian drugs for the duration of the trial.
12. The subject must be willing to participate in all study related activities and visits.

Exclusion Criteria:

1. Subjects who have had prior brain surgery.
2. Subjects with other major illnesses that could be complicated by amantadine exposure, including glaucoma, current hallucinations, urinary retention.
3. Subjects with dementia, depression and psychosis as determined by clinical examination.

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2010-01; Primary Completion 2012-04 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher G Goetz, MD, Principal Investigator — Rush University Medical Center; Glenn T Stebbins, PhD, Principal Investigator — Rush University Medical Center
Locations (8):
- United States (5):
  - University of Alabama-Birmingham (UAB), Birmingham, Alabama
  - University of South Florida, Tampa, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Duke University, Durham, North Carolina
  - Oregon Health & Science University (OHSU), Portland, Oregon
- Universitatsklinik fur Neurologie, Innsbruck, Austria
- Toronto Western Hospital (Movement Disorder Center), Toronto, Ontario, Canada
- Centre d'investigation Clinique, CHU de Toulouse, Toulouse, France

REFERENCES:
- See also: Parkinson's Disease Foundation — http://www.pdf.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Location: Medical clinics
Period: Overall Study
Arm/Group | Amantadine | Placebo
Started | 36 | 32
Completed | 31 | 30
Not Completed | 5 | 2
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Adverse Event | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Amantadine | Placebo | Total
Number analyzed (Participants) | 36 | 32 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.4 (8.2) | 68.5 (6.9) | 66.8 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 26 | 21 | 47
Region of Enrollment [Number; unit: participants]
  France | 2 | 4 | 6
  United States | 25 | 23 | 48
  Canada | 4 | 1 | 5
  Austria | 5 | 4 | 9
Movement Disorder Society revision of the Unified Parkinson's Disease Rating Scale MDS-UPDRS Part I [Mean (Standard Deviation); unit: units on a scale] — The Movement Disorder Society sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part I provides a measure of Non-Motor Experiences of Daily Living for the patient. These non-motor experiences include such items as cognitive function, psychosis and mood disturbances. Each item is rated on a 0 to 4 Likert type scale with 0 representing no impairment and 4 representing severe impairment. Part I score can range from 0 to 52.
  units on a scale | 9.8 (5.2) | 10.2 (5.2) | 10.0 (5.2)
MDS-UPDRS Part II [Mean (Standard Deviation); unit: units on a scale] — The Movement Disorder Society sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part II provides a measure of Motor Experiences of Daily Living for the patient using a Patient Reported Outcome approach. These motor experiences include such items as walking, fine motor or tremor disturbances. Each item is rated on a 0 to 4 Likert type scale with 0 representing no impairment and 4 representing severe impairment. Total Part II score can range from 0 to 52.
  units on a scale | 13.8 (5.8) | 14.3 (6.5) | 14.0 (6.1)
MDS-UPDRS Part III [Mean (Standard Deviation); unit: units on a scale] — The Movement Disorder Society sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III provides an objective (rater administered) measure of Parkinsonian motor impairment for the patient. These ratings are based on physical examination of the patient for signs such as tremor, rigidity, bradykinesia and postural instability. Each item is rated on a 0 to 4 Likert type scale with 0 representing no impairment and 4 representing severe impairment. Total Part III score can range from 0 to 132.
  units on a scale | 24.3 (10.7) | 20.3 (13.6) | 22.5 (12.2)
MDS-UPDRS Part IV [Mean (Standard Deviation); unit: units on a scale] — The Movement Disorder Society sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part IV provides a measure of complications of anti-parkinsonian treatment for the patient. These complications include such items as dyskinesia and dystonia. Each item is rated on a 0 to 4 Likert type scale with 0 representing no impairment and 4 representing severe impairment. Total Part IV score can range from 0 to 24.
  units on a scale | 8.5 (3.1) | 9.9 (3.6) | 9.2 (3.4)
Hoehn & Yahr Stage [Median (Full Range); unit: units on a scale] — The Hoehn and Yahr stage is a 0 to 5 Likert-type rating of global parkinsonian impairment with 0 representing no impairment and 5 representing inability to get out of bed or a wheelchair.
  units on a scale | 2 [1 to 4] | 2 [1 to 4] | 2 [1 to 4]

OUTCOME MEASURES:

1. Primary Outcome: The Investigators Will Assess Effect Size With Each Scale for Detecting Change From Baseline and Change Between Amantadine and Placebo; Allowing Assessment of Sensitivity and Specificity for Each Scale Based on Receiver Operator Characteristics (ROC).
Description: Analyses of primary outcome measures tested sensitivity to change in dyskinesia (time effect) as well as sensitivity to differences in treatment effect (time-by-treatment interaction). These analyses were conducted using repeated-measures ANOVA (RM-ANOVA) or nonparametric analyses (Friedman's ANOVA with follow-up Wilcoxon tests). The RM-ANOVAs tested for changes in scale scores over baseline, week 4, and week 8 visits across the entire sample (time effect), as well as differences in these changes over time between treatment groups (time-by-treatment interaction). Effect size of time to change was compared using a partial eta-square estimate of effect size. An eta-squared less than or equal to 0.01 is considered small; 0.06 is considered medium; and, 0.14 is considered large.
Time Frame: 18 months
Measure: Number; unit: unitless
Groups:
- Placebo: Placebo: Sugar pill given daily in three divided doses
Arm/Group | Amantadine | Placebo
Number analyzed (Participants) | 31 | 30
unitless | 0.061 | 0.061

ADVERSE EVENTS:
Time Frame: Adverse event recording occurred throughout the study duration.
Arm/Group | Amantadine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/32
Other Adverse Events (participants affected / at risk) | 4/36 | 3/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amantadine (N=36) | Placebo (N=32)
Dry mouth (Gastrointestinal disorders) | 4 (4) | 3 (3)

LIMITATIONS AND CAVEATS:
Study limitations include the patient population universally derived from university centers and the short duration of the program.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No